CLINICAL TRIAL: NCT02013674
Title: A Phase II, Randomized, Blinded, Study of the Safety and Efficacy of Transendocardial Injection of Allogeneic Human Mesenchymal Stem Cells (hMSCs) (20 Million or 100 Million Total MSCs) in Patients With Chronic Ischemic Left Ventricular Dysfunction Secondary to Myocardial Infarction.
Brief Title: The TRansendocardial Stem Cell Injection Delivery Effects on Neomyogenesis STudy (The TRIDENT Study)
Acronym: Trident
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Chief Science Officer, Director of Interdisciplinary Stem Cell Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120660
Record Dates: First submitted 2013-12-02; First posted 2013-12-17 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Ischemic Left Ventricular Dysfunction; Myocardial Infarction
Keywords: Cardiovascular; Chronic Ischemic Left Ventricular Dysfunction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: 20 million Allogeneic hMSCs (Experimental): Fifteen (15) patients to be treated with Allo-hMSCs: 4 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 0.2x 10^8 (20 million) Allo-hMSCs.
  Interventions: Biological: Allogeneic hMSCs
- Group 2: 100 million Allogeneic hMSCs (Experimental): Fifteen (15) patients to be treated with Allo-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1x 10^8 (100 million) Allo-hMSCs.
  Interventions: Biological: Allogeneic hMSCs

INTERVENTIONS:
Biological: Allogeneic hMSCs — Allogeneic Adult Human Mesenchymal Stem Cells (MSCs) delivered via injection
  Other Names: Allogeneic Adult Human Mesenchymal Stem Cells (MSCs)

SUMMARY:
Thirty (30) patients with chronic ischemic left ventricular dysfunction secondary to MI scheduled to undergo cardiac catheterization will be enrolled in the study. This is a phase II study intended to gain additional safety and efficacy assessments among two dose levels previously studied in a phase I setting.

DETAILED DESCRIPTION:
Thirty (30) patients with chronic ischemic left ventricular dysfunction secondary to MI scheduled to undergo cardiac catheterization will be enrolled in the study.This is a phase II study intended to gain additional safety and efficacy assessments among two dose levels previously studied in a phase I setting. In this study, a 20 million total hMSC dose and a 100 million total hMSC dose will be randomly allocated administered via the Biocardia Helical infusion system in a blinded manner.

The technique of transplanting progenitor cells into a region of damaged myocardium, termed cellular cardiomyoplasty, is a potentially new therapeutic modality designed to replace or repair necrotic, scarred, or dysfunctional myocardium. Ideally, graft cells should be readily available, easy to culture to ensure adequate quantities for transplantation, and able to survive in host myocardium, which is often a hostile environment of limited blood supply and immunorejection. Whether effective cellular regenerative strategies require that administered cells differentiate into adult cardiomyocytes and couple electromechanically with the surrounding myocardium is increasingly controversial and recent evidence suggests that this may not be required for effective cardiac repair. Most importantly, transplantation of graft cells should improve cardiac function and prevent adverse ventricular remodeling. To date, a number of candidate cells have been transplanted in experimental models, including fetal and neonatal cardiomyocytes, embryonic stem cell-derived myocytes, tissue engineered contractile grafts9, skeletal myoblasts, several cell types derived from adult bone marrow, and cardiac precursors residing within the heart itself. There has been substantial clinical development in the use of whole bone marrow and skeletal myoblast preparations in studies enrolling both post-infarction patients and patients with chronic ischemic left ventricular dysfunction and heart failure. The effects of bone marrow-derived mesenchymal stem cells (MSCs) have also been studied clinically.

Currently, bone marrow or bone marrow-derived cells represent a highly promising modality for cardiac repair. The totality of evidence from trials investigating autologous whole bone marrow infusions into patients following myocardial infarction supports the safety of this approach. In terms of efficacy, increases in ejection fraction are reported in the majority of the trials.

Chronic ischemic left ventricular dysfunction is a common and problematic condition; definitive therapy in the form of heart transplantation is available to only a tiny minority of eligible patients. Cellular cardiomyoplasty for chronic heart failure has been studied less than for acute MI, but represents a potentially important alternative for this disease.

ELIGIBILITY:
Inclusion Criteria:

* In order to participate in this study, a patient MUST:

  1. Be ≥ 21 and < 90 years of age.
  2. Provide written informed consent.
  3. Have a diagnosis of chronic ischemic left ventricular dysfunction secondary to myocardial infarction (MI) as defined by previous myocardial infarction documented by an imaging study demonstrating coronary artery disease with corresponding areas of akinesis, dyskinesis, or severe hypokinesis.
  4. Been treated with appropriate maximal medical therapy for heart failure or post-infarction left ventricular dysfunction. For beta-blockade, the patient must have been on a stable dose of a clinically appropriate beta-blocker for 3 months. For angiotensin-converting enzyme inhibition, the patient must have been on a stable dose of a clinically appropriate agent for 1 month.
  5. Be a candidate for cardiac catheterization within 5 to 10 weeks of screening as determined by doctors.
  6. Have an ejection fraction of less than or equal to 50% by gated blood pool scan, two-dimensional echocardiogram, CT, or left ventriculogram within the prior six months and not in the setting of a recent ischemic event.

Exclusion Criteria:

* In order to participate in this study, a patient MUST NOT:

  1. Have a baseline glomerular filtration rate ≤ 35 ml/min/1.73m2.
  2. Have a known, serious radiographic contrast allergy.
  3. Have a Mechanical aortic valve or heart constrictive device.
  4. Have a documented presence of aortic stenosis (aortic stenosis graded as 1.5cm2 or less).
  5. Have a documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥+2).
  6. Require coronary artery revascularization. Patients who require or undergo revascularization procedures should undergo these procedures a minimum of 3 months in advance of treatment in this study. In addition, patients who develop a need for revascularization following enrollment will be submitted for this therapy without delay.
  7. Have evidence of a life-threatening arrhythmia in the absence of a defibrillator (non-sustained ventricular tachycardia ≥ 20 consecutive beats or complete second or third degree heart block in the absence of a functioning pacemaker) or Corrected for heart rate (QTc) interval > 550 ms on screening ECG
  8. Automatic Implantable Cardioverter Defibrillator (AICD) firing in the past 60 days prior to enrollment.
  9. Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/µl or platelet values < 100,000/µl without another explanation.
  10. Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the upper limit of normal (ULN).
  11. Have a coagulopathy = (INR > 1.3) not due to a reversible cause (i.e., Coumadin). Patients on Coumadin will be withdrawn 5 days before the procedure and confirmed to have an INR < 1.3. Patients who cannot be withdrawn from Coumadin will be excluded from enrollment
  12. Have known allergies to penicillin or streptomycin.
  13. Hypersensitivity to Dimethyl Sulfoxide (DMSO).
  14. Be an organ transplant recipient.
  15. Have a history of organ or cell transplant rejection
  16. Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma.
  17. Have a non-cardiac condition that limits lifespan to < 1 year.
  18. Have a history of drug or alcohol abuse within the past 24 months.
  19. Be on chronic therapy with immunosuppressant medication, such as corticosteroids or TNFα antagonists.
  20. Be serum positive for HIV, hepatitis BsAg or viremic hepatitis C.
  21. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
  22. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI / University of Miami Miller School of Medicine
Locations (1):
- ISCI / University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Florea V, Rieger AC, DiFede DL, El-Khorazaty J, Natsumeda M, Banerjee MN, Tompkins BA, Khan A, Schulman IH, Landin AM, Mushtaq M, Golpanian S, Lowery MH, Byrnes JJ, Hendel RC, Cohen MG, Valasaki K, Pujol MV, Ghersin E, Miki R, Delgado C, Abuzeid F, Vidro-Casiano M, Saltzman RG, DaFonseca D, Caceres LV, Ramdas KN, Mendizabal A, Heldman AW, Mitrani RD, Hare JM. Dose Comparison Study of Allogeneic Mesenchymal Stem Cells in Patients With Ischemic Cardiomyopathy (The TRIDENT Study). Circ Res. 2017 Nov 10;121(11):1279-1290. doi: 10.1161/CIRCRESAHA.117.311827. Epub 2017 Sep 18. PMID 28923793
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School of Medicine — http://isci.med.miami.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (12.2) | 65.6 (9.4) | 66.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Enrollment Ejection Fraction (%) [Mean (Standard Deviation); unit: percentage] | 31.5 (9.9) | 26.7 (6.5) | 29.1 (8.6)
Enrollment Glomerular Filtration Rate (mL/Min) [Mean (Standard Deviation); unit: mL/min] | 70.0 (24.4) | 79.2 (20.4) | 74.6 (22.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAE).
Description: Incidence (at one month post-catheterization) of any treatment-emergent serious adverse events, defined as the composite of: death, non-fatal MI, stroke, hospitalization for worsening heart failure, cardiac perforation, pericardial tamponade, sustained ventricular arrhythmias (characterized by ventricular arrhythmias lasting longer than 15 seconds or with hemodynamic compromise).
Time Frame: One month post-catheterization
Population: SAEs are collected for 12 months, however, outcome 1 is only for SAEs during the first month.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

2. Secondary Outcome: Infarct Scar Size (ISS)
Description: Determined by delayed contrast enhanced Computed Tomography (CT) Scan
Time Frame: Baseline, 12 months
Population: Not all participants were able to complete procedure.
Measure: Median (Inter-Quartile Range); unit: Percent of Left Ventricular Mass
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Percent of Left Ventricular Mass
  Baseline | 9.9 [6.5 to 16.6] | 9.7 [6.5 to 12.3]
  12 Months: number analyzed (Participants) | 12 | 13
  12 Months | 6.8 [4.5 to 8.6] | 5.6 [4.7 to 6.9]

3. Secondary Outcome: Number of Participant With Reported Tissue Perfusion
Description: Tissue perfusion measured by CT.
Time Frame: 6 months, 12 months
Population: Not all participants were able to complete procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Participants
  at 6 months | 0 | 0
  at 12 months: number analyzed (Participants) | 12 | 13
  at 12 months | 0 | 0

4. Secondary Outcome: Peak Oxygen Consumption (VO2)
Description: Peak VO2 assessed via treadmill determination.
Time Frame: Baseline, 6 months, 12 months
Population: Not all participants were able to complete procedure.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
mL/kg/min
  Baseline | 15.8 (5.15) | 16.7 (4.48)
  6 months: number analyzed (Participants) | 14 | 12
  6 months | 15.0 (5.27) | 16.5 (5.30)
  12 months: number analyzed (Participants) | 13 | 14
  12 months | 14.4 (4.94) | 16.3 (5.84)

5. Secondary Outcome: Six-minute Walk Test.
Description: A test that measures how far a patient can walk in 6 minutes.
Time Frame: Baseline, 3 months, 6 months, 12 months
Population: Not all participants were able to complete procedure.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Meters
  Baseline | 398.7 (111.62) | 434.9 (120.04)
  3 months: number analyzed (Participants) | 14 | 15
  3 months | 396.1 (109.62) | 433.5 (133.97)
  6 months: number analyzed (Participants) | 14 | 14
  6 months | 416.4 (107.76) | 453.6 (126.82)
  12 months: number analyzed (Participants) | 14 | 14
  12 months | 409.7 (130.19) | 463.0 (143.07)

6. Secondary Outcome: Changed in New York Heart Association (NYHA) Functional Classification Based on Patient's Self Reported Activity Level.
Description: Changed in NYHA Functional Classification will be evaluated. Worsened: Documented increase in limitation in physical activity. Improved: Documented decrease in limitation in physical activity. Unchanged: No documented change in limitation in physical activity.
Time Frame: Baseline to 3 months, Baseline to 6 months, Baseline to 12 months
Population: Not all participants were able to complete procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Participants
  Baseline to 3 months, Improved | 2 | 4
  Baseline to 3 months, Unchanged | 10 | 9
  Baseline to 3 months, Worsened | 3 | 2
  Baseline to 6 months, Improved: number analyzed (Participants) | 14 | 14
  Baseline to 6 months, Improved | 5 | 4
  Baseline to 6 months, Unchanged: number analyzed (Participants) | 14 | 14
  Baseline to 6 months, Unchanged | 7 | 8
  Baseline to 6 months, Worsened: number analyzed (Participants) | 14 | 14
  Baseline to 6 months, Worsened | 2 | 2
  Baseline to 12 months, Improved: number analyzed (Participants) | 14 | 14
  Baseline to 12 months, Improved | 5 | 6
  Baseline to 12 months, Unchanged: number analyzed (Participants) | 14 | 14
  Baseline to 12 months, Unchanged | 8 | 4
  Baseline to 12 months, Worsened: number analyzed (Participants) | 14 | 14
  Baseline to 12 months, Worsened | 1 | 4

7. Secondary Outcome: Number of Incidents of Major Adverse Cardiac Events (MACE).
Description: Incidence of the Major Adverse Cardiac Events (MACE) endpoint, defined as the composite incidence of (1) death, (2) hospitalization for worsening heart failure, or (3) non-fatal recurrent MI.
Time Frame: 1 month, 6 months, 12 months post injection.
Population: Not all participants were able to complete study.
Measure: Number; unit: Incidents
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Incidents
  1 month from injection | 0 | 0
  6 months from injection | 3 | 2
  12 months from injection: number analyzed (Participants) | 14 | 14
  12 months from injection | 3 | 2

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (AE)
Description: Incidence of Treatment Emergent Adverse Event defined as any untoward medical occurrence in a patient or clinical investigation subject temporally associated with the use of the study product.
Time Frame: 6 months, 12 months
Population: Not all participants were able to complete the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Participants
  Treatment emergent AE (6 month) | 8 | 10
  Treatment emergent AE (12 months): number analyzed (Participants) | 14 | 14
  Treatment emergent AE (12 months) | 10 | 13

9. Secondary Outcome: Minnesota Living With Heart Failure (MLHF) Questionnaire Scores
Description: Minnesota Living with Heart Failure (MLHF) Questionnaire has a total score from 0 to 105. A higher score indicates that participant's heart failure is preventing them from living their life.
Time Frame: Baseline, 3 months, 6 months, 12 months
Population: Not all participants were able to complete procedure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 29.0 [21.0 to 52.0] | 35.0 [6.0 to 60.0]
  3 months | 22.0 [10.0 to 51.0] | 20.0 [6.0 to 40.0]
  6 months: number analyzed (Participants) | 15 | 14
  6 months | 30.0 [16.0 to 53.0] | 21.5 [9.0 to 34.0]
  12 months: number analyzed (Participants) | 14 | 14
  12 months | 25.0 [4.0 to 41.0] | 15.0 [8.0 to 64.0]

10. Secondary Outcome: Echocardiographic-derived Measures of Left Ventricular Function
Description: Left ventricular end diastolic wall thickness as determined by echocardiogram.
Time Frame: 6 months, 12 months
Population: Not all participants were able to complete the procedure.
Measure: Median (Inter-Quartile Range); unit: centimeters (cm)
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
centimeters (cm)
  Month 6: number analyzed (Participants) | 15 | 14
  Month 6 | 5.8 [5.2 to 6.3] | 6.3 [5.7 to 6.6]
  Month 12: number analyzed (Participants) | 14 | 13
  Month 12 | 6.1 [5.4 to 6.9] | 6.2 [5.4 to 6.6]

11. Secondary Outcome: Difference Between Regional Left Ventricular Function (at the Site of Allogeneic Cell Injections)
Description: As determined by Computed Tomography Scan
Time Frame: Baseline, 12 Months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Difference Between the Regional Left Ventricular Wall Thickening
Description: As determined by Computed Tomography Scan
Time Frame: Baseline, Month 12
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Difference Between Left Ventricular End Diastolic Wall Thickness
Description: As determined by Computed Tomography Scan
Time Frame: Baseline, 12 Months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Difference Between the Left Ventricular Ejection Fraction (LVEF)
Description: Change in 1-year LVEF by CT as compared to baseline.
Time Frame: Baseline, 12 months
Population: Not all participants were able to complete the procedure.
Measure: Median (Full Range); unit: Percentage of ejected blood
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 12 | 13
Percentage of ejected blood | -0.27 [-12.25 to 32.17] | 3.00 [-8.27 to 10.33]

15. Secondary Outcome: Difference in LVEF
Description: As assessed via ECHO
Time Frame: Baseline, 6 months, 12 months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Difference in Left Ventricular Volume
Description: Difference in left ventricular end diastolic and end systolic volume will be assessed via ECHO
Time Frame: Baseline, 6 months, 12 months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Difference in Left Ventricular Volume
Description: Difference in left ventricular end diastolic and end systolic volume will be assessed via CT
Time Frame: Baseline, 12 months
Population: Not all participants were able to complete the procedure.
Measure: Median (Full Range); unit: ml
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 12 | 13
ml | 7.65 [-15.89 to 44.76] | 3.70 [-43.85 to 53.66]

18. Secondary Outcome: Difference in Left Ventricular Regional Myocardial Perfusion
Description: As measured via myocardial mass by CT
Time Frame: Baseline, 12 months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Reads.
Description: The number of participants with abnormal ECG readings via 24 hour ambulatory ECG recordings as assessed per treating physician discretion.
Time Frame: 12 months
Population: Not all participants were able to complete the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
Participants
  baseline, normal | 0 | 1
  baseline, abnormal not clinically significant | 15 | 14
  baseline, abnormal, clinically significant | 0 | 0
  12 months, normal: number analyzed (Participants) | 12 | 14
  12 months, normal | 0 | 0
  12 months, abnormal not clinically significant: number analyzed (Participants) | 12 | 14
  12 months, abnormal not clinically significant | 12 | 14
  12 months, abnormal, clinically significant: number analyzed (Participants) | 12 | 14
  12 months, abnormal, clinically significant | 0 | 0

20. Secondary Outcome: Number of Clinically Significant of Abnormal Lab Values.
Description: Clinical significance of abnormal lab values will be assessed by treating physician
Time Frame: 12 months
Population: Data were not available to perform the statistical analyses as described in the protocol for this outcome.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Serial Troponin I
Description: Serial Troponin I values in ng/mL over time.
Time Frame: 12 hours, 24 hours post cardiac catheterization
Population: Not all participants were able to complete the procedure.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
ng/ml
  12-hours post-catheterization: number analyzed (Participants) | 14 | 13
  12-hours post-catheterization | 0.01 [0.01 to 0.10] | 0.01 [0.01 to 0.03]
  24-hours post-catheterization | 0.06 [0.01 to 0.29] | 0.05 [0.01 to 0.18]

22. Secondary Outcome: Number of Participants With Abnormal ECHO Reading
Description: The number of participants with abnormal reading post-cardiac catheterization. As assessed per treating physician discretion.
Time Frame: 6 hours post cardiac catheterization
Population: Not all participants were able to complete the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 7 | 8
Participants
  Normal | 1 | 2
  Abnormal, Not Clinically Significant | 6 | 6
  Abnormal, Clinically Significant | 0 | 0

23. Secondary Outcome: Creatinine Kinase Muscle/Brain (CK-MB)
Description: CK-MB values in ng/mL over time.
Time Frame: 12 hours, 24 hours post cardiac catheterization
Population: Not all participants were able to complete the procedure.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
Number analyzed (Participants) | 15 | 15
ng/ml
  12 hour post catheterization: number analyzed (Participants) | 14 | 14
  12 hour post catheterization | 3.25 [1.50 to 27.30] | 2.45 [1.20 to 6.20]
  24 hour post catheterization | 4.20 [2.40 to 19.30] | 4.40 [2.40 to 11.10]

ADVERSE EVENTS:
Time Frame: Adverse events are collected over approximately 1 year period.
Description: TE-SAE will only be reported for outcome 1 through 1 month post catheterization.
Arm/Group | Group 1: 20 Million Allogeneic hMSCs | Group 2: 100 Million Allogeneic hMSCs
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 4/15 | 2/15
Other Adverse Events (participants affected / at risk) | 8/15 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 20 Million Allogeneic hMSCs (N=15) | Group 2: 100 Million Allogeneic hMSCs (N=15)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) — Serious adverse events within 6 months of injection for acute coronary syndrome
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) — Serious adverse events within 6 months of injection
cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1) — Serious adverse events within 6 months of injection
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Serious adverse events within 6 months of injection
Arterisolerosis (Vascular disorders) | 0 (0) | 1 (1) — Serious adverse events within 6 months of injection
Haematoma (Vascular disorders) | 1 (1) | 0 (0) — Serious adverse events within 6 months of injection
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Serious adverse events within 6 months of injection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 20 Million Allogeneic hMSCs (N=15) | Group 2: 100 Million Allogeneic hMSCs (N=15)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Cardiac failure (Cardiac disorders) | 4 (4) | 0 (0) — Adverse events within 12 months of injection
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2) — Adverse events within 12 months of injection
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Sinus Arrest (Cardiac disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Eye Swelling (Eye disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Vision blurred (Eye disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Fatigue (General disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Gait disturbance (General disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Pyrexia (General disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Prostatic specific antigen (Investigations) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2) — Adverse events within 12 months of injection
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Adverse events within 12 months of injection
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) — Adverse events within 12 months of injection
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) — Adverse events within 12 months of injection
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Adverse events within 12 months of injection
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Stasis dematitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Haematoma (Vascular disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Chest Pain (General disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0) — Adverse events within 12 months of injection
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Impantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Adverse events within 12 months of injection
Spinal column ste (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Adverse events within 12 months of injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02013674/Prot_SAP_000.pdf